CLINICAL TRIAL: NCT04277481
Title: The Acute Effect of Cold Pack Therapy Applied on Healthy People for Different Periods on the Mechanical Properties of the Quadriceps Muscle
Brief Title: The Acute Effect of Cold Pack Therapy Applied on Healthy People for Different Periods
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Acibadem University (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-17/19
Record Dates: First submitted 2020-02-07; First posted 2020-02-20 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Cold; Muscle Injury
Keywords: Cold pack; Muscle
MeSH Terms: conditions — Common Cold

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1 (10 minute cold pack): 10 min, s package (35 * 29 cm) will be wrapped with a towel and applied to the rectus femoris part of the quadriceps.
  Interventions: Other: 10 minute cold pack
- Group 2 (12 minute cold pack): 12 min, s package (35 * 29 cm) will be wrapped with a towel and applied to the rectus femoris part of the quadriceps.
  Interventions: Other: 12 minute cold pack
- Group 3 (15 minute cold pack): 15 min, s package (35 * 29 cm) will be wrapped with a towel and applied to the rectus femoris part of the quadriceps.
  Interventions: Other: 15 minute cold pack
- Group 4 (20 minute cold pack): 20 min, s package (35 * 29 cm) will be wrapped with a towel and applied to the rectus femoris part of the quadriceps.
  Interventions: Other: 20 minute cold pack

INTERVENTIONS:
Other: 10 minute cold pack — 10 min package (35 * 29 cm) will be wrapped with a towel and applied to the rectus femoris part of the quadriceps.
  Groups: Group 1 (10 minute cold pack)
Other: 12 minute cold pack — 12 min package (35 * 29 cm) will be wrapped with a towel and applied to the rectus femoris part of the quadriceps.
  Groups: Group 2 (12 minute cold pack)
Other: 15 minute cold pack — 15, min package (35 * 29 cm) will be wrapped with a towel and applied to the rectus femoris part of the quadriceps.
  Groups: Group 3 (15 minute cold pack)
Other: 20 minute cold pack — 20 min package (35 * 29 cm) will be wrapped with a towel and applied to the rectus femoris part of the quadriceps.
  Groups: Group 4 (20 minute cold pack)

SUMMARY:
The cold pack application, which is a special silicate gel impregnated with water in a soft rubber envelope, is frequently applied in the clinic. It has been shown in the literature that local cold application causes increased resistance to movement. It is also reported that the muscle can change its mechanical properties in a short time. However, the effect of the cooling package application applied in different periods on the mechanical properties of the muscle is unknown. Therefore, in the current study proposal, the investigators aim to investigate the acute effect (0 min, 5 min, 10 min, 15 min, 20 min and 30 min) of cold pack therapy applied on healthy individuals for different periods (10-12-15-20 minutes).

DETAILED DESCRIPTION:
Cold Packs (Cold Pack, CP); Slika gel packs are the most commonly used modalities in clinics. Special silicate gel impregnated with water in a soft rubber envelope is stored in coolers whose temperature is maintained between -12.2 ° C and 9.4 ° C . There are different sizes and shapes. Since it does not lose its softness when it is cooled, it adapts well to the folds of the body. By putting a towel between the skin and the package, a homogeneous cooling is tried to be achieved, hygiene is provided and it is easier to tolerate the feeling of extreme cold felt in the first contact of the cold package. It can be applied for a relatively long time without losing its cold due to its low conductivity. Significant increase in package temperature is seen from the 15th minute of the application. It is stated that it decreases the skin temperature up to 10 ° C and keeps it at 20 ° C-30 ° C for 3 hours depending on the room temperature. They can be used repeatedly by cooling .

Intensive cold application for 12-15 minutes is enough to reduce pain and muscle spasm . It has also been shown that a cold application over 30 minutes can cause cold bite and nerve problems . However, in practical applications, cold appears to vary between 15-30 minutes for pain, muscle spasm and edema . In a review made by Auley regarding cryotherapy treatments; ice application has been shown to be used in 5 to 85 minutes in many studies. They said that cold application does not have a specified frequency and duration, but repeated 10 minutes of cold application is effective. In addition, it has been reported that there is evidence of a slightly less drop from 10 minutes to 20 minutes while the temperature drops in the first 10 minutes .

In animal studies performed in vitro, although muscle tissue has reported high resistance to strain after cooling, direct mechanical responses to muscles in human studies There is only one study that evaluates. In this study carried out by Mustalampi et al., Parameter measurements indicating the mechanical properties of the muscle immediately after applying the cold pack applied locally to the quadriceps muscle for 20 minutes and after 15 minutes. As a result of the study, the muscle has become stiffer, less elastic in terms of mechanical properties and it has been shown that these changes do not completely recover after 15 minutes. It was not observed when it was reinstated after fifteen minutes.

In the light of this information, in the current study proposal; the investigators aim to investigate the acute effect (0 min, 5 min, 10 min, 15 min, 20 min and 30 min) of the cold pack therapy on the mechanical properties of the quadriceps muscle in healthy people for different periods (10-12-15-20 minutes).

ELIGIBILITY:
Inclusion Criteria:

* Volunteer student between the ages of 18-23 with a subcutaneous fold thickness of the quadriceps muscle between 5 mm and 15 mm.
* Non-smoker
* No drug use

Exclusion Criteria:

Having any cardiovascular or peripheral vascular disease

* Known neuromuscular pathology history
* Having diabetes mellitus disease
* Having a history of lower limb pain and previous surgery
* Has a history of insensitivity to local heat or cold

Ages: 18 Years to 23 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Volunteer student between the ages of 18-23 with a subcutaneous fold thickness of the quadriceps muscle between 5 mm and 15 mm.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-02-12 (Estimated); Primary Completion 2020-02-28 (Estimated); Study Completion 2020-03-15 (Estimated)

PRIMARY OUTCOMES:
Measurement of skin temperature | Change from Baseline skin temperature at 0 minute, 5 minute, 10 minute, 20 minute past- cold pack
  For thermal imaging, a 120-9-90 pixel resolution FLIR E5 camera thermal camera (FLIR Systems AB, Sweden) will be used, and Color Palette iron will be selected to display images. The video will be taken from a distance of 1 m at a speed of 8 photos / s.
Evaluation of the mechanical properties of the muscle-1 | Change from Baseline mechanical properties at 0 minute, 10 minute, 20 minute past- cold pack
  Viscoelastic stiffness [N/m] will be measured in MyotonPro 3 (MYO, Tallin, Estonia).
Evaluation of the mechanical properties of the muscle-2 | Change from Baseline mechanical properties at 0 minute, 10 minute, 20 minute past- cold pack
  Oscillation frequency (Hz) will be measured in MyotonPro 3 (MYO, Tallin, Estonia).
Evaluation of the mechanical properties of the muscle-3 | Change from Baseline mechanical properties at 0 minute, 10 minute, 20 minute past- cold pack
  Mechanical stiffness (N/m) will be measured in MyotonPro 3 (MYO, Tallin, Estonia).

CONTACTS AND LOCATIONS:
Locations (1):
- Acibadem University, Istanbul, Ataşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mac Auley DC. Ice therapy: how good is the evidence? Int J Sports Med. 2001 Jul;22(5):379-84. doi: 10.1055/s-2001-15656. PMID 11510876
- [Background] Bizzini M, Mannion AF. Reliability of a new, hand-held device for assessing skeletal muscle stiffness. Clin Biomech (Bristol). 2003 Jun;18(5):459-61. doi: 10.1016/s0268-0033(03)00042-1. PMID 12763442
- [Background] Bleakley C, McDonough S, MacAuley D. The use of ice in the treatment of acute soft-tissue injury: a systematic review of randomized controlled trials. Am J Sports Med. 2004 Jan-Feb;32(1):251-61. doi: 10.1177/0363546503260757. PMID 14754753
- [Background] Enwemeka CS, Allen C, Avila P, Bina J, Konrade J, Munns S. Soft tissue thermodynamics before, during, and after cold pack therapy. Med Sci Sports Exerc. 2002 Jan;34(1):45-50. doi: 10.1097/00005768-200201000-00008. PMID 11782646
- [Background] Mustalampi S, Ylinen J, Kautiainen H, Weir A, Hakkinen A. Acute effects of cold pack on mechanical properties of the quadriceps muscle in healthy subjects. Phys Ther Sport. 2012 Nov;13(4):265-9. doi: 10.1016/j.ptsp.2012.02.001. Epub 2012 Apr 23. PMID 23068904